CLINICAL TRIAL: NCT05494112
Title: A Sub-Chronic Evaluation of the Safety of Celastrol in Human Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Legend Labz, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: AMT-002-2022
Record Dates: First submitted 2022-08-08; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Safety
MeSH Terms: interventions — celastrol

STUDY DESIGN:
Intervention Model Description: healthy men and women volunteers, between 18 and 40 years of age, over a 90-day period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amount of Celastrol Administered (Experimental): Chronic evaluation of the same doses of Celastrol to each subject over 90-day period
  Interventions: Dietary Supplement: Celastrol

INTERVENTIONS:
Dietary Supplement: Celastrol — same dose of Celastrol will be given every day for a period of 90-days to all participants.
  Other Names: 24,25,26-trinoroleana-1(10),3,5,7- tetraen-29-oic acid; 34157-83-0

SUMMARY:
This is an open label safety study that will not be blinded or placebo controlled.

Purpose is to evaluate the safety of Celastrol in healthy men and women volunteers, between 18 and 40 years of age, over a 90-day period.

Celastrol is different than Cholesterol. Cholesterol is a risk for heart disease. Celastrol is a natural occurring compound extracted from the root of Tripterygium wilfordii, a herb used in Chinese medicine.

DETAILED DESCRIPTION:
Pre-study Visit A pre-study visit will occur approximately one week before the scheduled beginning of the study. At this time all nutritional supplements must be stopped. During this visit, the subjects will sign an Informed Consent, will provide a medical history and list their concurrent medications. They will have a physical exam and then have a blood sample taken and receive an EKG. Women of child-bearing age will provide a urine sample to test for pregnancy. The subjects will then have their eligibility assessed based on the inclusion/exclusion criteria.

Study Visit 1, Day 0 The subjects who meet the entrance criteria will arrive at the clinic at an appointed time, and will again have their concurrent medications reviewed. They will be assigned a unique study number and be given a vial of experimental product that contains the same number as the subject, and contains ten capsules of product. Each capsule will contain ~67 mg of Celastrol. Instructions on how and when to take the experimental product will be given to the subjects by the clinician. A log book or an electronic portal will be presented to each subject so that daily information, such as the day and time of product ingestion, and any self-perceived adverse events, will be recorded. Any self-perceived adverse events experienced prior to taking any product should be told to the clinician at this time.

The subjects will be instructed to bring their drug vials to every clinic visit so that compliance can be determined. Any subject who has less than an 80% compliance rate will be excused from the study.

Study Visit 2, Day 2 To test for any acute effects of the experimental product, the subjects will return to the clinic on day 2 of the study. A blood sample will be taken, the log-book and vial will be reviewed for compliance, concurrent medications and any self-perceived adverse events will be discussed. Their vials that were given on Study Day 1 will contain enough remaining experimental product capsules to support the study to Day 7. Three extra capsules will be provided in the event that the subject cannot return to the clinic on the exact day indicated.

Study Visit 3, Day 7 The subjects will return to the clinic on Day 7, and a blood sample will be taken. As before, the log-book and vial will be reviewed for compliance, and concurrent medications and any self-perceived adverse events will be discussed. A vial containing enough experimental product, plus three additional capsules, to last another 7 days will be given.

Study Visit 4, Day 14 The clinic visit on Day 14 will mimic the visit on Day 7. However, during this visit the subjects will also receive a physical exam with vital signs, and an EKG. A vial containing enough product to last until Day 28 (Visit 5), plus 5 additional capsules, will be given to each subject.

Study Visits 5 and 6, Days 28 and 58 The clinic visits on Days 28 and 58 will again mimic the visit on Day 7. No EKGs will be taken. On Day 28, vials containing enough product, plus 5 additional capsules, to last to day 58 (Visit 6) will be given to each subject.

Study Visit 7, Day 88 The final clinic visit will consist of a physical exam with vital signs, a blood sample, and an EKG. The logbook and vial will be reviewed for compliance, and concurrent medications and any self-perceived adverse events will be discussed. At this point the study is complete and the subjects are released.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are between 18 and 40 years of age and who are found to be healthy without any underlying medical conditions and are not taking any daily medications. This does not exclude patients who take drugs prn.
2. Individuals who have not be involved in other clinical trials during the last 45 days. However, individuals that participated in the Celastrol-Sperm Health study can enter the trial after a seven day "wash-out" period
3. Women of child-bearing age and ability who agree to abstain from sexual intercourse, or agree to use condoms or vaginal diaphragms or other devices designed to prevent pregnancy; or are taking hormonal medication designed to prevent pregnancy, during the entire course of the study.
4. Women with tubal ligations or other physical conditions that make it impossible to conceive.
5. Women who are not pregnant or breast-feeding.

Exclusion Criteria:

1. Individuals who have been involved in any other clinical trial during the last 45 days.
2. Women of child-bearing age who do not agree to abstain from sexual intercourse, or do not agree to use condoms or vaginal diaphragms or other devices designed to prevent pregnancy, or who are not on hormonal medication designed to prevent pregnancy, during the entire course of the study.
3. Women who are pregnant or breast-feeding
4. Clinically significant cardiac disease including uncontrolled congestive heart failure and unstable angina
5. Individuals on medications that the clinician feels may interfere with the results
6. Medications that might interfere with blood chemistry, CBCs, or vital signs.
7. Subjects who are taking daily medications. The use of therapies prn, such as headache and allergy medication are allowed.
8. Subjects Less than 18 years of age
9. Prisoners
10. Subjects who have taken anabolic steroid use during the last six months.
11. Subjects with a current history of addictive alcohol or illegal drug abuse (e.g. cocaine, heroin, etc.). The use of marijuana is allowed.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-05-25 (Estimated); Study Completion 2023-05-25 (Estimated)

PRIMARY OUTCOMES:
The effect of celastrol on the function of the liver | 90 days
  Absence of Toxicity, as determined by comparison of periodic subject data to their baseline data

SECONDARY OUTCOMES:
EKG evaluation | 90 days
  Compared to laboratory standards
Glucose (MG/DL) | 90 days
  Glucose levels measured in the blood
BUN (MG/DL) | 90 days
  BUN levels measured in the blood
Creatine (MG/DL) | 90 days
  Creatine levels measured in the blood
eGFR (ML/MIN/1.73) | 90 days
  eGFR levels measured in the blood
CALC BUN/CREAT (Ratio) | 90 days
  Ratio of CALC BUN/CREAT measured in the blood
Sodium (MEQ/L) | 90 days
  Sodium levels measured in the blood
Potassium (MEQ/L) | 90 days
  Potassium levels measured in the blood
Chloride (MEQ/L) | 90 days
  Chloride levels measured in the blood
Carbon Dioxide (MEQ/L) | 90 days
  Carbon Dioxide levels measured in the blood
Calcium (MG/DL) | 90 days
  Calcium levels measured in the blood
Protein, Total (G/DL) | 90 days
  Total Protein levels measured in the blood
Albumin (G/DL) | 90 days
  Albumin levels measured in the blood
CALC Globulin (G/DL) | 90 days
  CALC Globulin levels measured in the blood
CALC A/G (Ratio) | 90 days
  Ratio of CALC A/G levels measured in the blood
Bilirubin, Total (MG/DL) | 90 days
  Bilirubin levels measured in the blood
Alkaline Phosphatase (U/L) | 90 days
  Alkaline Phosphatase levels measured in the blood
AST (U/L) | 90 days
  AST levels measured in the blood
ALT (U/L) | 90 days
  ALT levels measured in the blood
WBC (K/UL) | 90 days
  WBC levels measured in the blood
RBC (M/UL) | 90 days
  RBC levels measured in the blood
Hemoglobin (G/DL) | 90 days
  Hemoglobin levels measured in the blood
Hematocrit (%) | 90 days
  Hematocrit levels measured in the blood
MCV (fL) | 90 days
  MCV levels measured in the blood
MCH (PG) | 90 days
  MCH levels measured in the blood
MCHC (G/DL) | 90 days
  MCHC levels measured in the blood
RDW (%) | 90 days
  RDW levels measured in the blood
Neutrophils (%) | 90 days
  Neutrophils levels measured in the blood
Lymphocytes (%) | 90 days
  Lymphocytes levels measured in the blood
Monocytes (%) | 90 days
  Monocytes levels measured in the blood
Eosinophils (%) | 90 days
  Eosinophils levels measured in the blood
Basophils (%) | 90 days
  Basophils levels measured in the blood
Immature Granulocytes (%) | 90 days
  Immature Granulocytes levels measured in the blood
Nucleated RBCS (/100 WBC'S) | 90 days
  Nucleated RBCS levels measured in the blood
Platelet Count (K/UL) | 90 days
  Platelet Count levels measured in the blood
Absolute Neutrophils (K/UL) | 90 days
  Absolute Neutrophils levels measured in the blood
Absolute Monocytes (K/UL) | 90 days
  Absolute Monocytes levels measured in the blood
Absolute Eosinophils (K/UL) | 90 days
  Absolute Eosinophils levels measured in the blood
Absolute Basophils (K/UL) | 90 days
  Absolute Basophils levels measured in the blood
Absolute Immature Granulocytes (K/UL) | 90 days
  Absolute Immature Granulocyte levels measured in the blood
Absolute Nucleated RBCS (K/UL) | 90 days
  Absolute Nucleated RBCS levels measured in the blood
MPV (fL) | 90 days
  MPV levels measured in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Rubin Patel, MD, Principal Investigator — Patient Plus Urgent Care
Locations (1):
- Patient Plus Urgent Care, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Averages of collective patient data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: All data available on clinicaltrials.gov

REFERENCES:
- [Background] Kusy S, Ghosn EE, Herzenberg LA, Contag CH. Development of B cells and erythrocytes is specifically impaired by the drug celastrol in mice. PLoS One. 2012;7(4):e35733. doi: 10.1371/journal.pone.0035733. Epub 2012 Apr 24. PMID 22545133
- [Background] Hou W, Liu B, Xu H. Celastrol: Progresses in structure-modifications, structure-activity relationships, pharmacology and toxicology. Eur J Med Chem. 2020 Mar 1;189:112081. doi: 10.1016/j.ejmech.2020.112081. Epub 2020 Jan 20. PMID 31991334
- [Background] Sun H, Liu X, Xiong Q, Shikano S, Li M. Chronic inhibition of cardiac Kir2.1 and HERG potassium channels by celastrol with dual effects on both ion conductivity and protein trafficking. J Biol Chem. 2006 Mar 3;281(9):5877-84. doi: 10.1074/jbc.M600072200. Epub 2006 Jan 11. PMID 16407206
- [Background] Sun M, Tang Y, Ding T, Liu M, Wang X. Inhibitory effects of celastrol on rat liver cytochrome P450 1A2, 2C11, 2D6, 2E1 and 3A2 activity. Fitoterapia. 2014 Jan;92:1-8. doi: 10.1016/j.fitote.2013.10.004. Epub 2013 Oct 19. PMID 24144799
- [Background] Wang S, Liu K, Wang X, He Q, Chen X. Toxic effects of celastrol on embryonic development of zebrafish (Danio rerio). Drug Chem Toxicol. 2011 Jan;34(1):61-5. doi: 10.3109/01480545.2010.494664. Epub 2010 Oct 18. PMID 20954803
- [Background] Yuan YY, Gu ZP, Shi QX, Qin GW, Xu RS, Cao L. [In vitro inhibition of celastrol on spermatozoa fertilization ability of guinea pig]. Yao Xue Xue Bao. 1995;30(5):331-5. Chinese. PMID 7660802
- [Background] Zhang YS, Tu YY, Gao XC, Yuan J, Li G, Wang L, Deng JP, Wang Q, Ma RM. Strong inhibition of celastrol towards UDP-glucuronosyl transferase (UGT) 1A6 and 2B7 indicating potential risk of UGT-based herb-drug interaction. Molecules. 2012 Jun 5;17(6):6832-9. doi: 10.3390/molecules17066832. PMID 22669039